CLINICAL TRIAL: NCT01299467
Title: A Randomized, Double-Blind, Third Party Open, Double-Dummy, Placebo-Controlled, 3-Way Crossover Study To Determine The Duration Of Action Of Inhaled Doses Of PF-03526299 On Allergen-Induced Airway Responses In Mild Asthmatic Subjects
Brief Title: A Study To Assess The Duration Of Action Of PF-03526299 In Asthmatic Subjects Following Allergen Challenge
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: A9291006
Record Dates: First submitted 2011-01-03; First posted 2011-02-18 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: Asthma; duration of action; allergen challenge
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose 1 (0.5 hours) (Experimental)
  Interventions: Drug: Active (PF-03526299)
- Dose 1 (8 hours) (Experimental)
  Interventions: Drug: Active (PF-03526299)
- Dose 1 (placebo) (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose 2 (0.5 hr) (Experimental)
  Interventions: Drug: Active (PF-03526299)
- Dose 2 (8 hours) (Experimental)
  Interventions: Drug: Active (PF-03526299)
- Dose 2 (placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active (PF-03526299) — Capsules for inhalation, 1.396 mg twice a day for up to 13 days. Last dose given 0.5 hrs before allergen challenge
  Arms: Dose 1 (0.5 hours)
Drug: Active (PF-03526299) — Capsules for inhalation, 1.396 mg twice a day for up to 12 days. Last dose given 8 hrs before allergen challenge
  Arms: Dose 1 (8 hours)
Drug: Placebo — Capsules for inhalation, Placebo, twice a day for up to 13 days. Last dose given 0.5 hrs before allergen challenge
  Arms: Dose 1 (placebo)
Drug: Active (PF-03526299) — Capsules for inhalation, 4.188 mg twice a day for up to 13 days. Last dose given 0.5 hrs before allergen challenge
  Arms: Dose 2 (0.5 hr)
Drug: Active (PF-03526299) — Capsules for inhalation, 4.188 mg twice a day for up to 12 days. Last dose given 8hrs before allergen challenge
  Arms: Dose 2 (8 hours)
Drug: Placebo — Capsules for inhalation, Placebo, twice a day for up to 13 days. Last dose given 0.5 hrs before allergen challenge
  Arms: Dose 2 (placebo)

SUMMARY:
The purpose of this study is to find out how long the effect of PF-03526299 last after it is inhaled by assessing the lung function of mild asthma patients after they have been exposed to allergen

DETAILED DESCRIPTION:
To assess duration of action of the compound in suppressing the early and late allergen response in asthma patients

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 18 and 60 years, inclusive.
* A history or diagnosis of asthma that requires the use of beta 2 agonist bronchodilators (eg Salbutamol).
* Women who could become pregnant must use appropriate birth control throughout the study and pregnancy tests must be negative on entering the study and prior to dosing in the clinic.

Exclusion Criteria:

* Subjects who have been hospitalized for the treatment of asthma within three months prior to study entry, or have been hospitalized more than twice in last 12 months.
* Subjects who have experienced a lower respiratory tract infection (eg bronchitis or pneumonia) or significant asthma instability in the 4 weeks prior to study entry.
* Severe additional disease other than asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
To determine whether inhaled PF-03526299 has a sustained duration of action, using allergen-induced EAR in mild allergic asthmatics as a biomarker of response. | Up to 13 days

SECONDARY OUTCOMES:
To determine the effect of inhaled PF-03526299 after multiple dosing on allergen-induced EAR in mild allergic asthmatics. | Up to 13 days
To determine whether inhaled PF-03526299 has a sustained duration of action, using allergen-induced LAR in mild allergic asthmatics as a biomarker of response. | Up to 13 days
To investigate the safety, toleration and pharmacokinetics of an inhaled dose of PF-03526299 | Up ro 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9291006&StudyName=A%20Study%20To%20Assess%20The%20Duration%20Of%20Action%20Of%20PF-03526299%20In%20Asthmatic%20Subjects%20Following%20Allergen%20Challenge